CLINICAL TRIAL: NCT02162056
Title: Coronary and Structural Interventions Ulm - Bioresorbable Vascular Scaffold
Acronym: CSI-Ulm-BVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Jochen Wohrle, Prof. Dr. Jochen Wöhrle, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSI-Ulm-BVS 1.0
Record Dates: First submitted 2014-06-07; First posted 2014-06-12 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Stable Angina; Unstable Angina; Acute Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Angina, Stable; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- use of bioresorbable vascular scaffolds (Experimental): Implantation of bioresorbable vascular scaffold for coronary artery disease.
  Interventions: Device: use of bioresorbable vascular scaffolds

INTERVENTIONS:
Device: use of bioresorbable vascular scaffolds — Implantation of bioresorbable vascular scaffolds for coronary artery disease.

SUMMARY:
To evaluate the safety, performance and efficacy of the bioresorbable vascular scaffold (BVS) system in patients with coronary artery disease

DETAILED DESCRIPTION:
Patients with coronary artery disease receive bioabsorbable vascular scaffolds. Patients are clinically followed during a period of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease
* implantation of at least one bioresorbable vascular scaffold

Exclusion Criteria:

* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2013-11; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wöhrle, MD, Principal Investigator — University of Ulm, Ulm, Germany
Locations (1):
- University of Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reichart C, Wohrle J, Markovic S, Rottbauer W, Seeger J. Clinical results of bioresorbable drug-eluting scaffolds in short and long coronary artery lesions using the PSP technique. BMC Cardiovasc Disord. 2019 Jan 18;19(1):22. doi: 10.1186/s12872-018-0994-y. PMID 30658574
- [Derived] Markovic S, Kugler C, Rottbauer W, Wohrle J. Long-term clinical results of bioresorbable absorb scaffolds using the PSP-technique in patients with and without diabetes. J Interv Cardiol. 2017 Aug;30(4):325-330. doi: 10.1111/joic.12392. Epub 2017 Jun 1. PMID 28568564
- [Derived] Markovic S, Dragomir S, Walcher D, Bernhardt P, Imhof A, Rottbauer W, Wohrle J. Clinical results of single and multiple bioresorbable drug-eluting scaffolds for treatment of de-novo coronary artery disease. Coron Artery Dis. 2016 Nov;27(7):561-5. doi: 10.1097/MCA.0000000000000392. PMID 27244371